CLINICAL TRIAL: NCT02922985
Title: Multimodal Pain Management for Cesarean Delivery: A Randomized Control Trial
Brief Title: Multimodal Pain Management for Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB 16-0121
Record Dates: First submitted 2016-09-29; First posted 2016-10-04 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2017-10

CONDITIONS: Pain
Keywords: Cesarean delivery; Multimodal pain management
MeSH Terms: conditions — Pain | interventions — Acetaminophen; Ketorolac; Injections, Intramuscular; Ketorolac Tromethamine; Bupivacaine; Injections, Subcutaneous; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Control Group (Placebo Comparator): Patients will receive a placebo dose of all three study medications: Patients will receive the pre-operative dose of IV normal saline placebo within 30 minutes of going to the OR for CD. The patient will receive the subcutaneous infiltration of 20 mL of subcutaneous normal saline placebo after positioning and preparation but prior to skin incision. At the time of fascial closure, the patient will receive an IM dose of normal saline placebo.
  Interventions: Drug: Normal saline
- Multimodal Pain Regimen Group (Active Comparator): Patients will receive the actual study medication for all three study medications: Patients will receive the pre-operative dose of IV acetaminophen 1 g within 30 minutes of going to the OR for CD. The patient will receive the subcutaneous infiltration of either 20 mL of bupivacaine 0.25% after positioning and preparation but prior to skin incision. At the time of fascial closure, the patient will receive 60 mg of IM ketorolac.
  Interventions: Drug: Intravenous acetominophen; Drug: Ketorolac, intramuscular; Drug: Bupivacaine, subcutaneous

INTERVENTIONS:
Drug: Intravenous acetominophen — One dose if 1 gram intravenous to be given pre-surgery
  Other Names: Ofirmev
  Arms: Multimodal Pain Regimen Group
Drug: Ketorolac, intramuscular — One dose of 60 mg Intramuscular to be given at time of skin closure
  Other Names: Toradol
  Arms: Multimodal Pain Regimen Group
Drug: Bupivacaine, subcutaneous — Inject 20 mL of 0.25% bupivacaine at the site of anticipated skin incision.
  Arms: Multimodal Pain Regimen Group
Drug: Normal saline — Normal saline will be given intravenously, intra-muscularly, and subcutaneously in the same volume as the study drugs for the patients in the placebo group.
  Arms: Placebo Control Group

SUMMARY:
Opioid use and abuse has become a major medical problem in the United States. Over prescription of opioid medications is a major contributor to this growing problem. Cesarean delivery (CD) is the most commonly performed surgery in the US and women are generally given opioid medications for postoperative pain management. This is not a common practice in other developed countries. We believe that a multimodal pain management strategy is superior to current practices for control of postoperative pain after CD and will lead to a decrease in the use of opioid medications. This will have beneficial effects on patients' recovery and bonding with their newborns, as well as societal effects in reducing the burden of opioid abuse in the US. Our objective is to investigate the use of a multimodal pain regimen in pregnant patients undergoing CD. This is a randomized double-blinded, placebo controlled trial. The multimodal intervention consists of a pre-operative dose of IV acetaminophen (Ofirmev), infiltration of subcutaneous bupivacaine prior to skin incision, and a dose of IM ketorolac at time of fascial closure. These study medications are currently used in our patient population but not in a standardized fashion, not in every patient, and not always in combination with each other. The control group will receive placebo IV infusion preoperatively and an IM injection at fascial closure, and subcutaneous infiltration with normal saline before skin incision. Both groups will receive spinal regional anesthesia as per anesthesia team and then postoperatively, both groups will receive the current standard of care, which consists postoperative hydrocodone/acetaminophen and ibuprofen as needed depending on pain score. Our primary outcome of interest will be the total opioid intake in the first 48 hours after surgery. Secondary outcomes include time to first opioid given, pain scores at 6-12, 24 and 48 hours post op, and total number of opioid tablets left after discharge on post op day number 7. We will also evaluate patient satisfaction scores and total length of hospital stay. We will evaluate neonatal outcomes including Apgar scores, cord blood gases, immediate newborn complications in the first 48 hours after birth, and any infant adverse outcomes related to maternal opioid use up to 4 weeks of life. Our hypothesis is that our multimodal pain regimen will decrease the total opioid requirement in the first 48 hours after surgery.

DETAILED DESCRIPTION:
We are proposing a double-blinded, placebo controlled, randomized trial of patients undergoing elective cesarean delivery. Participants will be randomized to either a control group or study group. This is a double-blinded study, neither participants nor the obstetric or anesthesia team are aware of study assignment. The study group, aka multimodal group, will receive 1 g of IV acetaminophen (ofirmev) within 30 minutes before starting the surgery, regional anesthesia (spinal anesthesia only) with fentanyl, duramorph (morphine) and bupivacaine will be performed as per anesthesia team, the anticipated sight of skin incision will be infiltrated with 20 mL of bupivacaine 0.25% in the subcutaneous space prior to skin incision, and 60 mg of intramuscular (IM) ketorolac (toradol) will be given at the time of fascial closure. The control group will receive a placebo drip within 30 minutes before starting the surgery, regional anesthesia (spinal anesthesia only) with fentanyl, duramorph (morphine) and bupivacaine will be performed as per anesthesia team, the anticipated sight of skin incision will be infiltrated with 20 mL of normal saline in the subcutaneous space prior to skin incision, and an IM dose of placebo at the time of fascial closure. Post-operatively both groups will be managed similarly.

Inclusion Criteria:

* Women who are 18 - 45 years of age at the time of cesarean delivery with the ability to give informed consent
* Elective cesarean delivery
* Gestational age ≥ 34 weeks
* Fluent in either English or Spanish
* Spinal anesthesia

Exclusion Criteria:

Urgent or emergent CD Active labor Epidural or Intrathecal regional anesthesia General anesthesia Patients with a contraindication for regional anesthesia Acute or chronic hepatic disease Acute or chronic renal disease Active asthma Gastrointestinal ulceration Inflammatory bowel disease Allergy to ketorolac, acetaminophen, hydrocodone, codeine, ibuprofen or bupivacaine Opioid dependence Non reassuring fetal or maternal status requiring immediate delivery Placenta previa or accreta Acute or chronic pain disorder Maternal weight <50 kilograms Uncontrolled hypertension Ischemic cardiac disease Congestive heart failure Thrombocytopenia, platelet count <150,000/microliter Preeclampsia including Hemolysis Elevated Liver enzymes Low Platelets syndrome DIC or active hemorrhage before randomization Estimated blood loss > 2000 mL

Primary Outcome: The primary outcome of the study is the total opioid (hydrocodone) use in milligrams in the first 48 hours after cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Women who are 18 - 45 years of age at the time of cesarean delivery with the ability to give informed consent
* Elective cesarean delivery
* Gestational age ≥ 34 weeks
* Fluent in either English or Spanish
* Spinal anesthesia

Exclusion Criteria:

* Urgent or emergent CD
* Epidural or combined spinal epidural regional anesthesia
* General anesthesia
* Patients with a contraindication for regional anesthesia
* Acute or chronic hepatic disease
* Acute or chronic renal disease
* Active asthma
* Gastrointestinal ulceration
* Inflammatory bowel disease
* Allergy to ketorolac, acetaminophen, hydrocodone, codeine, ibuprofen or bupivacaine
* Opioid dependence
* Non reassuring fetal or maternal status requiring immediate delivery
* Placenta previa or accreta
* Acute or chronic pain disorder
* Maternal weight <50 kilograms
* Uncontrolled hypertension
* Ischemic cardiac disease
* Congestive heart failure
* Thrombocytopenia, platelet count <150,000/microliter
* Preeclampsia including Hemolysis Elevated Liver enzymes Low Platelets syndrome
* Disseminated intravascular coagulation (DIC) or active hemorrhage before randomization
* Estimated blood loss > 2000 mL

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2016-10; Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily E Hadley, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

REFERENCES:
- [Background] Bartels K, Mayes LM, Dingmann C, Bullard KJ, Hopfer CJ, Binswanger IA. Opioid Use and Storage Patterns by Patients after Hospital Discharge following Surgery. PLoS One. 2016 Jan 29;11(1):e0147972. doi: 10.1371/journal.pone.0147972. eCollection 2016. PMID 26824844
- [Background] Santoso JT, Ulm MA, Jennings PW, Wan JY. Multimodal pain control is associated with reduced hospital stay following open abdominal hysterectomy. Eur J Obstet Gynecol Reprod Biol. 2014 Dec;183:48-51. doi: 10.1016/j.ejogrb.2014.10.007. Epub 2014 Oct 14. PMID 25461352
- [Background] Rosaeg OP, Lui AC, Cicutti NJ, Bragg PR, Crossan ML, Krepski B. Peri-operative multimodal pain therapy for caesarean section: analgesia and fitness for discharge. Can J Anaesth. 1997 Aug;44(8):803-9. doi: 10.1007/BF03013154. PMID 9260006
- [Background] Munishankar B, Fettes P, Moore C, McLeod GA. A double-blind randomised controlled trial of paracetamol, diclofenac or the combination for pain relief after caesarean section. Int J Obstet Anesth. 2008 Jan;17(1):9-14. doi: 10.1016/j.ijoa.2007.06.006. Epub 2007 Nov 5. PMID 17981455
- [Derived] Hadley EE, Monsivais L, Pacheco L, Babazade R, Chiossi G, Ramirez Y, Ellis V, Simon M, Saade GR, Costantine M. Multimodal Pain Management for Cesarean Delivery: A Double-Blinded, Placebo-Controlled, Randomized Clinical Trial. Am J Perinatol. 2019 Sep;36(11):1097-1105. doi: 10.1055/s-0039-1681096. Epub 2019 Mar 1. PMID 30822800

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Control Group: Patients will receive a placebo dose of all three study medications
  Normal saline: Normal saline will be given intravenously, intra-muscularly, and subcutaneously in the same volume as the study drugs for the patients in the placebo group.
- Multimodal Pain Regimen Group: Patients will receive the actual study medication for all three study medications.
  Intravenous acetominophen: One dose if 1 gram intravenous to be given pre-surgery
  Ketorolac, intramuscular: One dose of 60 mg Intramuscular to be given at time of skin closure
  Bupivacaine, subcutaneous: Inject 20 mL of 0.25% bupivacaine at the site of anticipated skin incision.
Period: Overall Study
Arm/Group | Placebo Control Group | Multimodal Pain Regimen Group
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Control Group | Multimodal Pain Regimen Group | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 60 | 120
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (5.2) | 29.6 (5.1) | 29.5 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 60 | 120
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Hispanic | 39 | 40 | 79
  Race: Caucasian | 13 | 12 | 25
  Race: African American | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120
worst pain in the last 24 hours prior to cesarean delivery [Median (Inter-Quartile Range); unit: score on a scale] — patients report of the score of worst pain in the last 24 hours prior to cesarean delivery, expressed on a scale from 0-10. A higher score means worse pain (worse outcome).
  score on a scale | 2 [0 to 6] | 3 [0 to 6] | 2 [0 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Intake in Morphine Milligram Equivalents in the First 48 Hours After Cesarean Delivery (CD)
Description: Every opioid intake by the patient in the first 48 hours after CD will be recorded and quantified in morphine milligram equivalents
Time Frame: 48 hours post cesarean delivery
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalents
Arm/Group | Placebo Control Group | Multimodal Pain Regimen Group
Number analyzed (Participants) | 60 | 60
morphine milligram equivalents | 42 [30 to 60] | 49.5 [32 to 69]

2. Secondary Outcome: Time to First Administration of Opioid Pain Medication Post Operatively
Description: Time, in hours, to first administration of opioid pain medication post operatively
Time Frame: 48 hours post cesarean delivery
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Placebo Control Group | Multimodal Pain Regimen Group
Number analyzed (Participants) | 60 | 60
hours | 6.05 [1.9 to 13.5] | 6.35 [2.2 to 16.3]

3. Secondary Outcome: Pain Score at 6-12 Hours Post Operatively
Description: Pain score at 6-12 hours post-operatively, expressed on a pain scale from 0-10 with the higher score meaning worse pain (outcome).
Time Frame: 6-12 hours post-operatively
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo Control Group | Multimodal Pain Regimen Group
Number analyzed (Participants) | 60 | 60
score on a scale | 6 [2 to 7] | 6 [0.25 to 7]

4. Secondary Outcome: Number of Opioid Pain Tablets Remaining on Post-operative Day #7 From the Discharge Prescription.
Description: Number of opioid pain tablets remaining on post-operative day #7 from hospital discharge as reported by patients
Time Frame: 7 days post delivery
Population: We could not get the outcome on two patients from placebo control group and three patients from multimodal pain regimen group due to patients not responding to calls. These 5 five subjects were considered lost to follow up for this outcome.
Measure: Median (Inter-Quartile Range); unit: Tablets
Arm/Group | Placebo Control Group | Multimodal Pain Regimen Group
Number analyzed (Participants) | 58 | 57
Tablets | 18 [12 to 24] | 19 [8.5 to 25]

5. Secondary Outcome: Hospital Length of Stay
Description: Time to discharge from hospital, measured in hours
Time Frame: From time of hospital admission to time of discharge home up to 168 hours.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Placebo Control Group | Multimodal Pain Regimen Group
Number analyzed (Participants) | 60 | 60
hours | 50.2 [41.5 to 52.5] | 50 [42.9 to 52]

6. Secondary Outcome: Pain Score at 24 Hours Post-operatively
Description: Pain Score at 24 Hours Post Operatively, expressed on a pain scale from 0-10 with the higher score meaning worse pain (outcome).
Time Frame: 24 hours post-operatively
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo Control Group | Multimodal Pain Regimen Group
Number analyzed (Participants) | 60 | 60
score on a scale | 5 [2 to 7] | 6 [3 to 7]

7. Secondary Outcome: Pain Score at 48 Hours Post-operatively
Description: Pain Score at 48 Hours Post-operatively, expressed on a pain scale from 0-10 with the higher score meaning worse pain (outcome).
Time Frame: 48 hours post-operatively
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo Control Group | Multimodal Pain Regimen Group
Number analyzed (Participants) | 60 | 60
score on a scale | 4 [0 to 6] | 3 [0 to 6]

8. Secondary Outcome: Apgar Score at 5 Minutes
Description: This is the Apgar score of the newborn collected at 5 minutes. Range is from 0-10, with the higher scores meaning a better outcome.
Time Frame: 5 minutes after birth
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo Control Group | Multimodal Pain Regimen Group
Number analyzed (Participants) | 60 | 60
score on a scale | 9 [9 to 9] | 9 [9 to 9]

9. Secondary Outcome: NICU Admission
Description: Rate of admission to the neonatal intensive care unit
Time Frame: after birth and before hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Control Group | Multimodal Pain Regimen Group
Number analyzed (Participants) | 60 | 60
Participants | 2 | 6

10. Secondary Outcome: Need for Respiratory Support
Description: neonate receipt of oxygen by nasal cannula or mechanical ventilation
Time Frame: after birth and before hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Control Group | Multimodal Pain Regimen Group
Number analyzed (Participants) | 60 | 60
Participants | 0 | 4

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Placebo Control Group | Multimodal Pain Regimen Group
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 2/60 | 1/60
Other Adverse Events (participants affected / at risk) | 1/60 | 2/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Control Group (N=60) | Multimodal Pain Regimen Group (N=60)
October 2016-May 2017 (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) — Postpartum hemorrhage
October 2016-May 2018 (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — Fascial dehiscence
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Control Group (N=60) | Multimodal Pain Regimen Group (N=60)
October 2016-May 2017 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Severe skin itching
October 2016-May 2018 (Renal and urinary disorders) | 0 (0) | 1 (1) — Urinary retention
October 2016-May 2017 (Cardiac disorders) | 1 (1) | 0 (0) — Chest pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT02922985/Prot_SAP_000.pdf